CLINICAL TRIAL: NCT05408598
Title: Cognitive and Functional Trajectories in Older Adults After a Pharmacologic Multidisciplinary Intervention: a Study Protocol
Brief Title: Pharmacological Optimization by a Specialized Outpatient Consultation Team
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Principal Investigator, Nicolás Martínez Velilla, Head of Geriatric Unit, Fundacion Miguel Servet
Other Study IDs: PHARM-OPTIMIZ GERIATRÍA
Record Dates: First submitted 2022-03-01; First posted 2022-06-07 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-06

CONDITIONS: Polypharmacy
Keywords: Geriatrics; Pharmacist; Outpatient; Polypharmacy; Medication review; Functional capacity; Cognitive capacity; Comprehensive Geriatric Assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background Polypharmacy is a common condition among older adults and is a major issue of concern for its association with adverse drug reactions and adverse health outcomes, including falls, functional and cognitive impairment, frailty, and increased use of healthcare resources. Therefore, an appropriate interprofessional collaboration is essential to face this growing concern. In our outpatient clinic, we have initiated a new approach to provide specialized care for older adults based on a close collaboration between different professionals to optimize drug therapy. With the aim to assess the impact of this specialized outpatient clinic on patients' abilities, a prospective study will be conducted in community-dwelling older adults with polypharmacy.

Methods The present study will be conducted with geriatric outpatients with polypharmacy (defined as ≥ 5 prescribed medications at the time of inclusion) in the Navarra University Hospital, a Spanish Public tertiary University Hospital. At least 104 patients aged 75 years or older, with a life expectancy ≥ 3 months willing to provide informed consent will be recruited from the outpatient clinic. Drug optimization in the first consultation will be accompanied by subsequent face-to-face and/or telephone follow-up at intermediate (~ 3 months) and end of study (~ 6 months). The primary endpoint will be the change in functional and cognitive capacities measured at baseline and follow-up. Secondary endpoints will be the analysis of medication changes (i.e. number of medications and drugs, type of intervention, anticholinergic burden, and the number of STOPP/START criteria), change in patient's quality of life, rate of falling, and use of healthcare resources.

Discussion Regarding geriatric outpatients, studies in which medication review has been conducted by a multidisciplinary team (at least comprising a physician and a pharmacist) functional and cognitive patient's capacities have not been reported. What this study adds is the impact of a specialized consultation team focused on pharmacotherapy optimization in functional and cognitive abilities of community-dwelling older adults with polypharmacy. A multidisciplinary approach to polypharmacy could be an effective way for improving patients' functional and cognitive abilities. We expect that the association of different complementary professional roles working together will have a synergistic effect and will be an effective strategy for this purpose.

ELIGIBILITY:
Inclusion criteria:

* ≥ 75 years old
* Willing to provide informed consent
* Life expectancy ≥ 3 months
* Present polypharmacy (defined as ≥ 5 prescribed medications at the time of inclusion).

Exclusion Criteria:

* Refusal to sign the informed consent form by the patient/primary caregiver/legal guardian or inability to obtain it.
* Participation in a clinical trial related to medication.
* In the event of a no-show or cancellation of the appointment at the first visit.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community-dwelling older adults ( ≥ 75 years old) with polypharmacy (defined as ≥ 5 prescribed medications at the time of inclusion).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-11-20 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in functional capacity: Barthel Index (spanish version) | 12 months
  The change in Barthel Index measured at baseline and follow-up (measure of Basic Activities of Daily Living)
Change in functional capacity: Lawton Scale (spanish version) | 12 months
  The change in Lawton Scale measured at baseline and follow-up (measure of Instrumental Activities of Daily Living)
Change in functional capacity: Short Physical Performance Battery test (SPPB; Spanish versión) | 12 months
  The change in SPPB measured at baseline and follow-up (measure of balance, gait, and rising from a chair)
Change in functional capacity: Strenght (Handgrip) | 12 months
  The change in Strenght measured at baseline and follow-up
Change in cognitive function by the "Índice de Incapacidad psíquica de la Cruz Roja" (IPCR). | 12 months
  The change in IPCR measured at baseline and follow-up

SECONDARY OUTCOMES:
Quality of life (changes between baseline and follow-up) | 12 months
  Quality of life, assessed by the questionnaire EQ-5D-5L (Spanish version) and a subjectively rated visual analog scale (EQ VAS).
Frailty(changes between baseline and follow-up) | 12 months
  Frailty will be assessed by Fried criteria and Frail-VIG.
Healthcare use | 12 months
  Comparison of healthcare use (hospital admissions, primary care and emergency visits) between baseline and follow-up consultations.
Burden of medications between baseline and follow-up. | 12 months
  The analysis of medication changes between baseline and follow-up will comprise: number of medications and drugs, anticholinergic burden assessed by drug burden index (DBI) and Anticholinergic Burden Calculator (ACB) scales, and number of STOPP/START criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Navarra (HUN), Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share data under reasonable request

REFERENCES:
- [Derived] Roncal-Belzunce V, Gutierrez-Valencia M, Cedeno-Veloz BA, San Miguel R, Marin-Epelde I, Galbete A, Preciado Goldaracena J, Ezpeleta MI, Garaioa-Aramburu K, Martinez-Velilla N. Impact of a Multidisciplinary Approach to Polypharmacy Management in Community-Dwelling Older Adults: Insights From a Specialized Outpatient Clinic. Aging Med (Milton). 2025 Feb 18;8(1):e70001. doi: 10.1002/agm2.70001. eCollection 2025 Feb. PMID 39968007
- [Derived] Roncal-Belzunce V, Cedeno-Veloz BA, Elcano RSM, Gutierrez-Valencia M, Izquieta VR, Guruceaga-Eguillor I, Marin-Epelde I, Echeverria-Beistegui I, Sanchez-Latorre M, Galbete A, Garaioa-Aramburu K, Martinez-Velilla N. Cognitive and functional trajectories in geriatric outpatients after a pharmacologic multidisciplinary intervention: A study protocol. Rev Esp Geriatr Gerontol. 2023 Sep-Oct;58(5):101386. doi: 10.1016/j.regg.2023.101386. Epub 2023 Jul 29. PMID 37523939